CLINICAL TRIAL: NCT03062267
Title: Effectiveness of a Mobile Texting Intervention for People With Serious Mental Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Dror Ben-Zeev, Professor, School of Medicine: Psychiatry and Behavioral Sciences, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00001274
Record Dates: First submitted 2017-02-09; First posted 2017-02-23 (Actual); Results first posted 2020-11-09 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-10

CONDITIONS: Schizoaffective Disorder; Schizophrenia; Bipolar Disorder; Major Depressive Disorder
Keywords: mhealth; texting intervention; mobile health; mobile mental health
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia; Bipolar Disorder; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as Usual (No Intervention): Treatment as usual for 3 months.
- Mobile Interventionist (Experimental): Participants will exchange text messages with a mobile interventionist throughout the day for 3 months.
  Interventions: Other: Mobile Interventionist

INTERVENTIONS:
Other: Mobile Interventionist — A mobile interventionist is a trained clinician who provides supportive messaging through text messages via mobile devices (i.e. basic / smartphones)
  Arms: Mobile Interventionist

SUMMARY:
Testing an mHealth mobile interventionist texting program on illness management.

DETAILED DESCRIPTION:
The ultimate objective is to evaluate a validated mHealth intervention that can be realistically integrated into community mental health settings to increase the availability, reach, and broad impact of illness management approaches for people with serious mental illness (SMI).

ELIGIBILITY:
Inclusion Criteria:

1. Chart diagnosis of schizophrenia, schizoaffective disorder, bipolar disorder, or major depressive disorder;
2. 18 years or older;
3. A rating of "3" or higher on one of three Patient Activation items;
4. Ownership of a mobile phone with call/text plan (research staff will offer assistance in accessing the Federal Lifeline Assistance Program to people who do not have a mobile phone and/or call/text plan if they are otherwise eligible);
5. Receiving community based treatment services.

Exclusion Criteria:

1. Hearing, vision, or motor impairment that make it impossible to operate a mobile phone (determined using the individual's device for screening);
2. English reading level below 4th grade (determined using the reading section from the Wide Range Achievement Test - 4th Edition (WRAT-4).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dror Ben-Zeev, PhD, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - Thresholds, Chicago, Illinois
  - Frontier Behavioral Health, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No significant events to report that occurred after participant enrollment but prior to assignment of participants to an arm.
Period: Overall Study
Arm/Group | Treatment as Usual | Mobile Interventionist
Started | 12 | 37
Completed | 10 | 32
Not Completed | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment as Usual | Mobile Interventionist | Total
Number analyzed (Participants) | 12 | 37 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (12.0) | 45.4 (11.1) | 44.8 (11.2)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 7 | 15 | 22
  Male | 5 | 22 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 9 | 33 | 42
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 10 | 12
  White | 7 | 17 | 24
  More than one race | 2 | 6 | 8
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 12 | 37 | 49

OUTCOME MEASURES:

1. Primary Outcome: Psychiatric Symptoms
Description: Assessed with the Psychotic Symptom Rating Scales (PSYRATS). The PSYRATS inquires about the specific dimensions of hallucinations and delusions. There are 17 items and each item is rated from 0 (absent) to 4 (severe). The PSYRATS has 2 subscales: the auditory hallucinations subscale (AHS) consisting of 11 items, and the delusions subscale (DS) consisting of 6 items. These subscale scores are added to create a total score ranging from 0-68. Higher scores indicate worse symptoms.
Time Frame: Change from baseline to 3 months and 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment as Usual | Mobile Interventionist
Number analyzed (Participants) | 12 | 37
score on a scale
  Score at Baseline | 5.2 (11.2) | 19.6 (20.4)
  Score at 3 months | 6.2 (14.4) | 15.1 (16.7)
  Score at 6 months | .6 (1.9) | 17.9 (19.1)

2. Primary Outcome: Psychiatric Symptoms
Description: Assessed with the Beck Depression Inventory (BDI). The Beck Depression Inventory is a psychometric test for measuring the severity of depression. There are 21 items, each rated from 0-3, and total scores range from 0-63. Higher scores indicate more severe depressive symptoms.
Time Frame: Change from baseline to 3 months and 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment as Usual | Mobile Interventionist
Number analyzed (Participants) | 12 | 37
score on a scale
  Score at Baseline | 18.5 (13.7) | 18.5 (11.4)
  Score at 3 Months | 17.2 (11.3) | 23.4 (12.4)
  Score at 6 Months | 15.5 (11.2) | 14.8 (10.3)

3. Secondary Outcome: Recovery
Description: Assessed with the Recovery Assessment Scale (RAS). This scale measures mental health recovery. There are 24 items, each rated from 1 (disagree) to 5 (agree), and total scores range from 24-120. Higher scores indicate better recovery.
Time Frame: Change from baseline to 3 months and 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment as Usual | Mobile Interventionist
Number analyzed (Participants) | 12 | 37
score on a scale
  Score at Baseline | 91.8 (14.6) | 89.8 (17.3)
  Score at 3 Months | 90.0 (13.8) | 92.9 (15.5)
  Score at 6 Months | 93.8 (13.1) | 94.4 (14.9)

4. Other Pre Specified Outcome: Satisfaction With Treatment
Description: Assessed with satisfaction items established from previous SMI research. This measure consists of 5 items, each rated from 1 (strongly disagree) to 7 (strongly agree), and total scores range from 5-35. Higher scores indicate more satisfaction with treatment.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment as Usual | Mobile Interventionist
Number analyzed (Participants) | 12 | 37
score on a scale | 28.2 (6.2) | 30.1 (6.1)

ADVERSE EVENTS:
Time Frame: 6 months.
Arm/Group | Treatment as Usual | Mobile Interventionist
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/37
Other Adverse Events (participants affected / at risk) | 0/12 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-09): https://cdn.clinicaltrials.gov/large-docs/67/NCT03062267/Prot_SAP_000.pdf